CLINICAL TRIAL: NCT03059550
Title: Screening for Glucose Metabolism Disorders in Cardiac Rehabilitation After an Acute Coronary Syndrome (REHABDIAB [REHABilitation for Coronary Disease and DIABetes])
Brief Title: Screening for Glucose Metabolism Disorders in Cardiac Rehabilitation
Acronym: REHABDIAB
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Principal Investigator, Prof. Bruno Vergès, Professor, Centre Hospitalier Universitaire Dijon
Other Study IDs: CHUDijon
Record Dates: First submitted 2017-02-16; First posted 2017-02-23 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Diabetes
Keywords: cardiac rehabilitation; prediabetes
MeSH Terms: conditions — Diabetes Mellitus; Prediabetic State

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cardiac rehabilitation: Patients reffered to cardiac Rehabilitation after an acute coronary syndrome
- Whole French population post-ACS: The whole French population who presented an acute coronary syndrome (ACS) in the years 2013 and 2014.

SUMMARY:
Because prevalence of glucose metabolism disorders is high in patients with coronary disease, the Oral Glucose Tolerance Test (OGTT) is recommended in all patients without diabetes after an acute coronary syndrome (ACS). However, there are some concerns about its performance in clinical practice. The aim of our study was to evaluate, after an acute coronary syndrome (ACS), the feasibility and efficacy of the OGTT in a cardiac rehabilitation (CR) center in comparison with its real application in the whole French population.

DETAILED DESCRIPTION:
We will select all the patients referred to our Cardiac Rehabilitation center after an ACS. HbA1c will be measured in each patient included in the study. the OGTT will be prescribed in all the patients without known diabetes and with HbA1c < 6.5%. In order to perform a "real life" study, the OGTT will not performed in the CR center but will prescribed in each patient who will be asked to perform it in an external biological laboratory.

The OGTT will be performed in the morning after a 12 hour fast, with 75g oral glucose load. Plasma glucose will be measured at baseline and 120 min after the oral glucose load. The results will be classified according to the WHO criteria: diabetes is defined as fasting plasma glucose (FPG) greater or equal to 7.0 mmol/L (126 mg/dL) or glucose level 2h (2hPG) after the OGTT greater or equal to 11.1mmol/L (200mg/dL); impaired fasting glucose (IFG) is defined as FPG greater or equal to 6.1 mmol/L (110mg/dL) and less than 7.0 mmol/L and impaired glucose tolerance (IGT) is defined as a 2hPG greater or equal to 7.8 mmol/L (140 mg/dL) and less than 11.1mmol/L.

In parallel, screening for glucose metabolism disorders with the OGTT after an ACS will be evaluated in the whole French population from a representative sample of 1/97ème French population of the "National Health Insurance Inter-Regime Information System" (SNIIRAM) which collects individual hospital and non-hospital data for health care consumption.

ELIGIBILITY:
Inclusion Criteria:

* patients referred to cardiac rehabilitation after an acute coronary syndrome during the 6 precious weeks

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients referred to cardiac rehabilitation after an acute coronary syndrome
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2013-03-01 (Actual); Primary Completion 2015-05-31 (Actual); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of OGTT performed after an acute coronary syndrome | 26 months
  Percentage of OGTT performed after an acute coronary syndrome

SECONDARY OUTCOMES:
Abnormalities of glucose metabolism diagnosed in cardiac rehabilitation | 26 months
  Abnormalities of glucose metabolism diagnosed in cardiac rehabilitation: diabetes, impaired glucose tolerance, impaired fasting glucose
Profile of the patients according to their glucose abnormalities | 26 months
  Clinical, biological and peak workload in each category of patients, normoglycemic, patients with diabetes, patients with impaired glucose tolerance, patients with impaired fasting glucose

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Vergès, MD, PhD, Principal Investigator — CHU Dijon
Locations (1):
- CHU Dijon, Dijon, Burgundy, France

IPD SHARING:
Plan to Share IPD: Undecided